CLINICAL TRIAL: NCT06107803
Title: A Phase 1b, In-Patient Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of the Co-Administration of Roluperidone and Olanzapine in Adult Subjects With Moderate to Severe Negative Symptoms of Schizophrenia
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Co-Administration of Roluperidone and Olanzapine in Adult Subjects With Moderate to Severe Negative Symptoms of Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minerva Neurosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MIN-101C18
Record Dates: First submitted 2023-10-13; First posted 2023-10-30 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Negative Symptoms in Schizophrenia
MeSH Terms: interventions — roluperidone; Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Phase 1 (Experimental): Roluperidone 64 mg monotherapy administered as an oral dose daily for 7 days on Days 1-7.
  Interventions: Drug: Roluperidone 64 mg
- Treatment Phase 2 (Experimental): Roluperidone 64 mg oral and olanzapine 10 mg oral administered at the same time daily for 10 days on Days 8-17.
  Interventions: Drug: Roluperidone 64 mg; Drug: Olanzapine 10 MG

INTERVENTIONS:
Drug: Roluperidone 64 mg — 64 mg/day oral
  Other Names: MIN-101
Drug: Olanzapine 10 MG — 10 mg/day oral
  Arms: Treatment Phase 2

SUMMARY:
The goal of this clinical trial is to evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of the Co-Administration of Roluperidone and Olanzapine in Adult Subjects with Moderate to Severe Negative Symptoms of Schizophrenia.

The main question this clinical trial aims to answer are the pharmacodynamic and pharmacokinetic effects and safety of the concomitant therapy of Roluperidone with an established and widely used antipsychotic, such as olanzapine in order to provide further guidance to clinical practitioners that may prescribe off-label use of these drugs concomitantly in clinical practice.

Eligible Participants will undergo the following study phases in the clinic:

* Screening Phase: Between 2 and up to 28 days during which study eligibility will be established and subjects receiving psychotropics will be washed out. Subjects will remain inpatient at the clinical site at least through the end of Treatment Phase 2.
* Treatment Phase 1: After the Baseline Visit, Roluperidone 64 mg/day will be administered as a monotherapy for 7 days (Days 1-7).
* Treatment Phase 2: Concomitant administration of Olanzapine 10 mg/day and Roluperidone 64 mg/day for 10 days, starting on Day 8 (Days 8-17). Subjects may be discharged from the clinic at least 48 hours after the last administration of the study drugs and after the collection of the last plasma sample; however, the inpatient period may be extended at the discretion of the investigator.

End of Study (EOS): Will take place at least 14 days after the last dose of the study.

ELIGIBILITY:
Inclusion Criteria:

* Provided informed consent
* Body mass index (BMI) < 35 kg/m2
* Meets the diagnostic criteria for schizophrenia as defined in the Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-5), as established by a full psychiatric interview in conjunction with the Mini International Neuropsychiatric Interview (MINI)
* Documented diagnosis of schizophrenia for at least 1 year before screening
* Stable in terms of both positive and negative symptoms of schizophrenia over the last 3 months
* Score of > 20 on the PANSS original negative symptoms subscale (Sum of N1+N2+N3+N4+N5+N6+N7) at Screening and Baseline (Day -1) AND < 4 points absolute difference between the 2 visits
* Discontinued psychotropic medications without risk to their clinical status or safety by Baseline
* Female subject, if not of childbearing potential, must be a woman who is post-menopausal or permanently sterilized
* Female subject, if of childbearing potential, must test negative for pregnancy and must be using a double barrier contraceptive method
* Must be normal metabolizer for P450 CYP 2D6, defined as a subject that has at least one functional allele (eg, *1, *2 or *35), as determined by study-specific genotyping test before the first drug dose is administered
* Has a caregiver or family member or health care personnel who can provide information towards assessment and support the subject in terms of compliance with the protocol

Exclusion Criteria:

* Current major depressive disorder, bipolar disorder, panic disorder, obsessive compulsive disorder, or intellectual disability (intellectual developmental disorder diagnosed by age 14)
* PANSS item score of > 4 on:

  * P4 Excitement/Hyperactivity
  * P6 Suspiciousness/persecution
  * P7 Hostility
  * G8 Uncooperativeness
  * G14 Poor impulse control
* CDSS total score > 6
* Score of ≥ 2 on any 2 of items 1, 2, or 3, or a score of ≥ 3 on item 4 of the Barnes Akathisia Rating Scale (BARS)
* Has had electroconvulsive therapy (ECT), vagal nerve stimulation (VNS), or repetitive trans-cranial magnetic stimulation (r-TMS) within the 6 months prior to the Screening visit or who are scheduled for ECT, VNS, or r-TMS at any time during the study
* Positive urine drug screen for drugs of abuse
* Currently taking proton pump inhibitors (PPI)
* Current systemic infection (eg, Hepatitis B, Hepatitis C, human immunodeficiency virus [HIV], tuberculosis)
* Requires or may require concomitant treatment with any other medication likely to increase QT interval
* Requires medication inhibiting CYP2D6
* Safety laboratory results show one or more of the following: potassium <3.4 mmol/L, or calcium <2.07 mmol/L, or magnesium <0.70 mmol/L

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Collaborative Neuroscience Research, LLC, Garden Grove, California
  - CBH Health, LLC, Gaithersburg, Maryland
  - Hassman Research Institute, Marlton, New Jersey

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent three study phases: Screening, Treatment Phase 1 and Treatment Phase 2.
Groups:
- Overall Safety Set: 17 subjects were enrolled and received ≥ 1 dose of study drug and were included in the Safety Set.
Period: Overall Study
Arm/Group | Overall Safety Set
Started | 17
Full Set | 17
Safety Set | 17
Pharmacokinetic Set | 12
Pharmacokinetic Completer Set | 11
Completed | 13
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall Safety Set
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Body Mass Index at Baseline [Mean (Standard Deviation); unit: kg/m2] | 27.3 (4.58)

OUTCOME MEASURES:

1. Primary Outcome: Extrapyramidal Symptoms Assessed by Abnormal Involuntary Movement Scale (AIMS) - Change From Baseline in AIMS Component Movement
Description: AIMS is a rating scale to measure tardive dyskinesia (TD). For the scoring, the AIMS scale has 14 items. The first 10 items (under categories of Facial and Oral Movements, Extremity Movements, Trunk Movements, and Global Judgements) are rated from 0 (none) to 4 (severe); the remaining 4 items (Dental Status) are rated "yes" and "no" and not counted. The analysis is limited to items 1 to 10, with each rated from 0 to 4. The total score is the sum of all 10 items and with values ranging from 0 to 40. Overall change from baseline to End of Study (Day 17) in AIMS was reported for the Safety Set. Higher scores imply worse outcome.
Time Frame: Overall - Change from Baseline to End of Study (Day 17)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Safety Set
Number analyzed (Participants) | 17
score on a scale | 0.0 (0.00)

2. Primary Outcome: Barnes Akathisia Rating Scale (BARS)
Description: BARS is a multiple-choice questionnaire that clinicians may use to provide an assessment of akathisia. The clinician or rater is instructed to observe the subject while standing and while sitting, at least 2 minutes each (total of at least 4 minutes in total). There are 4 areas where the subject is to be evaluated, 1 of these is objective, 2 are subjective, and the final is a global assessment. The BARS scale has 3 items that are rated from 0 (absence/no distress) to 3 (most severe). The BARS rating scale is scored by summing the scales for Objective Akathisia, Subjective Awareness of Restlessness and Subjective Distress Related to Restlessness yielding a total score ranging from 0 to 9. The Total score, which has a possible range from 0-9, is reported. Higher scores imply worse outcome.
Time Frame: Overall - Change from Baseline to End of Study (Day 17)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Safety Set
Number analyzed (Participants) | 17
score on a scale | 0.0 (0.00)

3. Primary Outcome: Number of Subjects Who Experienced Suicidal Ideation or Behavior Events Per the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a measure to identify and assess individuals at risk for suicide. Questions are phrased for an interview format but can be completed as a self-report measure if needed. It measures 4 constructs: severity of ideation, intensity of ideation, behavior, and lethality. It includes "stem questions," which if endorsed, prompt additional follow-up questions to obtain more information. For the composite endpoint of suicidal ideation or behavior (1-10), the number and percent of subjects in the Overall Safety Set who experience any one of the ten suicidal ideation or behavior events at End of Study (Day 17).
Time Frame: Overall - End of Study (Day 17)
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Safety Set
Number analyzed (Participants) | 17
Participants | 0

4. Secondary Outcome: Pharmacokinetic Evaluation of Roluperidone - Maximum Plasma Concentration (Cmax)
Description: Cmax of roluperidone and its metabolite following single dose and at steady state, and when administered concomitantly with olanzapine.
Time Frame: Days 1 through 17
Population: Treatment Phase 1 - Day 7 had 15 participants analyzed. Treatment Phase 2 - Day 17 had 13 participants analyzed.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Overall Safety Set - Roluperidone; Overall Safety Set - Metabolite BFB-520: Roluperidone 64 mg monotherapy administered as an oral dose daily for 7 days on Days 1-7 and concomitantly with olanzapine 10 mg daily on Days 8-17.
Arm/Group | Overall Safety Set - Roluperidone | Overall Safety Set - Metabolite BFB-520
Number analyzed (Participants) | 17 | 17
ng/ml
  Treatment Phase 1 - Day 1 | 32.5 (13.7) | 5.00 (5.69)
  Treatment Phase 1 - Day 7: number analyzed (Participants) | 15 | 15
  Treatment Phase 1 - Day 7 | 43.6 (19.9) | 7.98 (6.78)
  Treatment Phase 2 - Day 17: number analyzed (Participants) | 13 | 13
  Treatment Phase 2 - Day 17 | 67.7 (28.6) | 12.2 (12.9)

5. Secondary Outcome: Pharmacokinetic Evaluation of Roluperidone - Time to Maximum Plasma Concentration (Tmax)
Description: Tmax of roluperidone and its metabolite following single dose and at steady state, and when administered concomitantly with olanzapine.
Time Frame: Days 1 through 17
Population: Treatment Phase 1 - Day 7 had 15 participants analyzed. Treatment Phase 2 - Day 17 had 13 participants analyzed.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Overall Safety Set - Roluperidone | Overall Safety Set - Metabolite BFB-520
Number analyzed (Participants) | 17 | 17
hr
  Treatment Phase 1 - Day 1 | 9.74 (7.37) | 16.2 (6.72)
  Treatment Phase 1 - Day 7: number analyzed (Participants) | 15 | 15
  Treatment Phase 1 - Day 7 | 7.47 (5.73) | 9.60 (6.02)
  Treatment Phase 2 - Day 17: number analyzed (Participants) | 13 | 13
  Treatment Phase 2 - Day 17 | 6.20 (4.56) | 8.76 (4.90)

6. Secondary Outcome: Pharmacokinetic Evaluation of Roluperidone - Area Under the Plasma Concentration Versus Time Curve (AUC 0-24)
Description: AUC of roluperidone and its metabolite following single dose and at steady state, and when administered concomitantly with olanzapine.
Time Frame: Days 1 through 17
Population: Treatment Phase 1 - Day 7 had 15 participants analyzed. Treatment Phase 2 - Day 17 had 13 participants analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Overall Safety Set - Roluperidone | Overall Safety Set - Metabolite BFB-520
Number analyzed (Participants) | 17 | 17
hr*ng/mL
  Treatment Phase 1 - Day 1 | 391 (252) | 52.3 (63.0)
  Treatment Phase 1 - Day 7: number analyzed (Participants) | 15 | 15
  Treatment Phase 1 - Day 7 | 507 (278) | 135 (122)
  Treatment Phase 2 - Day 17: number analyzed (Participants) | 13 | 13
  Treatment Phase 2 - Day 17 | 720 (321) | 203 (225)

7. Secondary Outcome: Pharmacokinetic Evaluation of Roluperidone - Area Under the Plasma Concentration Versus Time Curve (AUC Inf)
Description: as for outcome 6
Time Frame: Days 1 through 17
Population: Treatment Phase 1 - Day 7 had 15 participants analyzed. Treatment Phase 2 - Day 17 had 13 participants analyzed.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Overall Safety Set - Roluperidone | Overall Safety Set - Metabolite BFB-520
Number analyzed (Participants) | 17 | 17
hr*ng/mL
  Treatment Phase 1 - Day 1 | 338 (289) | 60.7 (82.0)
  Treatment Phase 1 - Day 7: number analyzed (Participants) | 15 | 15
  Treatment Phase 1 - Day 7 | 495 (272) | 168 (234)
  Treatment Phase 2 - Day 17: number analyzed (Participants) | 13 | 13
  Treatment Phase 2 - Day 17 | 883 (420) | 263 (280)

8. Secondary Outcome: Plasma PK Parameter for Olanzapine Cmax
Description: Cmax of olanzapine administered concomitantly with roluperidone
Time Frame: Treatment Phase 2 (Day 8 through Day 17)
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Treatment Phase 2 - Day 17: Roluperidone 64 mg + Olanzapine 10 mg
Arm/Group | Treatment Phase 2 - Day 17
Number analyzed (Participants) | 13
ng/ml | 35.6 (12.7)

9. Secondary Outcome: Plasma PK Parameter for Olanzapine Tmax
Description: Tmax of olanzapine administered concomitantly with roluperidone
Time Frame: Treatment Phase 2 (Day 8 through Day 17)
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment Phase 2 - Day 17
Number analyzed (Participants) | 13
hr | 4.11 (2.24)

10. Secondary Outcome: Plasma PK Parameter for Olanzapine AUC 0-24
Description: AUC 0-24 olanzapine administered concomitantly with roluperidone
Time Frame: Treatment Phase 2 (Day 8 through Day 17)
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Treatment Phase 2 - Day 17
Number analyzed (Participants) | 13
hr*ng/ml | 587 (220)

11. Secondary Outcome: Plasma PK Parameter for Olanzapine AUC Inf
Description: AUC inf olanzapine administered concomitantly with roluperidone
Time Frame: Treatment Phase 2 (Day 8 through Day 17)
Measure: Mean (Standard Deviation); unit: hr*ng/ml
Arm/Group | Treatment Phase 2 - Day 17
Number analyzed (Participants) | 13
hr*ng/ml | 719 (144)

12. Secondary Outcome: Pharmacokinetic Evaluation of Co-administration Versus Roluperidone Monotherapy - Maximum Plasma Concentration (Cmax)
Description: Comparison of roluperidone on Day 17 with olanzapine to roluperidone alone on Day 7 for Cmax.
  The geometric mean and geometric coefficient of variation are reported for the analytes roluperidone and its metabolite.
Time Frame: Days 1 through 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Reference - Roluperidone Alone on Day 7: Roluperidone 64 mg
- Test - Roluperidone With Olanzapine on Day 17: Roluperidone 64 mg + Olanzapine 10 mg
Arm/Group | Reference - Roluperidone Alone on Day 7 | Test - Roluperidone With Olanzapine on Day 17
Number analyzed (Participants) | 15 | 13
ng/ml
  Roluperidone Analyte | 39.8 (46.37) | 62.2 (44.78)
  BFB-520 Analyte | 5.96 (89.12) | 8.54 (100.10)

13. Secondary Outcome: Pharmacokinetic Evaluation of Co-administration - AUC 0-24
Description: Comparison of roluperidone on Day 17 with olanzapine to roluperidone alone on Day 7 for AUC 0-24.
  The geometric mean and geometric coefficient of variation are reported for the analytes roluperidone and its metabolite.
Time Frame: Days 1 through 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Reference - Roluperidone Alone on Day 7 | Test - Roluperidone With Olanzapine on Day 17
Number analyzed (Participants) | 15 | 13
hr*ng/ml
  Roluperidone Analyte | 451 (50.50) | 656 (48.37)
  BFB-520 Analyte | 95.7 (103.10) | 135 (107.95)

ADVERSE EVENTS:
Time Frame: Treatment through end of study (Day 17).
Arm/Group | Treatment Phase 1 | Treatment Phase 2
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/15
Other Adverse Events (participants affected / at risk) | 5/17 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Phase 1 (N=17) | Treatment Phase 2 (N=15)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Phase 1 (N=17) | Treatment Phase 2 (N=15)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT06107803/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT06107803/SAP_001.pdf